CLINICAL TRIAL: NCT03051646
Title: A Placebo-controlled Double Blind Crossover Trial of Acetylsalicylic Acid as a Pre-treatment for Exercise in Multiple Sclerosis
Brief Title: Aspirin as a Pre-Treatment for Exercise in Multiple Sclerosis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Victoria M. Leavitt, Assistant Professor of Neuropsychology, Columbia University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: AAAQ1758
Record Dates: First submitted 2017-02-08; First posted 2017-02-14 (Actual); Results first posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Fatigue; Overheating
Keywords: Exercise; Time to Exhaustion
MeSH Terms: conditions — Fatigue; Sunstroke; Motor Activity | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: Design is a within-subject crossover placebo-controlled experiment. Each participant will be seen for two exercise sessions (stationary cycling) on two days separated by one week, and will receive either ASA or placebo (treatment) at each session prior to commencing exercise. Order of treatment will be randomized and counter-balanced. As such, each participant will serve as his/her own control.
Who Masked: Participant, Investigator
Masking Description: Blinding will be overseen by the CUMC pharmacy; randomization schedule will be submitted to the pharmacy by a third party who is not involved in the study (i.e., non-study personnel). Study investigators will remain blinded until data collection is complete and data have been analyzed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- Acetylsalicylic acid first, placebo second (Experimental): Participant is administered acetylsalicylic acid one hour prior to exercise.
  Interventions: Drug: Acetylsalicylic acid at 1st visit, then Placebo at 2nd visit
- Placebo oral capsule first, ASA second (Placebo Comparator): Participant is administered placebo one hour prior to exercise.
  Interventions: Drug: Placebo at 1st visit, then Acetylsalicylic acid at 2nd visit

INTERVENTIONS:
Drug: Acetylsalicylic acid at 1st visit, then Placebo at 2nd visit — 650 mg dose of acetylsalicylic acid is administered in a capsule one hour prior to exercise; Placebo oral capsule is administered one hour prior to exercise
  Other Names: aspirin; placebo
  Arms: Acetylsalicylic acid first, placebo second
Drug: Placebo at 1st visit, then Acetylsalicylic acid at 2nd visit — Placebo oral capsule is administered one hour prior to exercise; 650 mg dose of acetylsalicylic acid is administered in a capsule one hour prior to exercise
  Other Names: placebo; aspirin
  Arms: Placebo oral capsule first, ASA second

SUMMARY:
Exercise has many benefits for people with multiple sclerosis (MS), such as improved physical symptoms, mood, fatigue, and cognition. However, many people with MS refrain from exercising because of the discomfort of exhaustion and overheating that they experience. This study investigates the use of aspirin before exercise as a treatment to reduce overheating and exhaustion, thereby availing many more people with MS the opportunity to benefit from exercise.

The investigators recently published the first-ever report of elevated body temperature in relapsing-remitting MS (RRMS) patients relative to healthy controls, and elevated temperature was linked to worse fatigue. This finding that body temperature is elevated and linked to fatigue in RRMS lays the groundwork for a paradigm shift in our understanding and treatment of fatigue. That is, the focus shifts from exogenous to endogenous temperature, and from stimulant medication to cooling treatments.

A recent study comparing healthy adults to adults with MS showed that whereas exercise increased body temperature in both groups, only in the MS group was it correlated with exhaustion. The reason for this may relate to the elevation in resting body temperature in relapsing-remitting MS (RRMS) patients relative to healthy controls. The finding is clinically meaningful, as elevated body temperature was correlated with worse fatigue in patients. Exercise Aim: To determine whether pretreatment with ASA (compared to placebo: within subject crossover design) before exercise results in improved exercise performance (i.e., increased time-to-exhaustion). The investigators hypothesize that participants will tolerate exercise for longer after taking ASA than placebo. This hypothesis is based on a) demonstrated efficacy of antipyretic for reducing body temperature during exercise in healthy controls, b) demonstrated efficacy of antipyretic for reducing fatigue in non-exercising MS patients, and c) demonstrated efficacy of elaborate (unblinded) cooling treatments (e.g., cooling garments, cooling hand chamber) for improving exercise performance in MS patients. Note that this project is especially important for MS patients, who have a disease-specific body temperature elevation and sensitivity to heat (i.e., Uhthoff's).

DETAILED DESCRIPTION:
Exercise is beneficial for people with MS. Exercise has many benefits for persons with multiple sclerosis (MS), including increased muscle strength, improved balance, decreased fatigue, decreased depression, improved memory, and improved quality of life. In addition to clinical improvements, there is direct and indirect neural evidence for beneficial effects of exercise in MS. For example, work in the experimental autoimmune encephalopathy (EAE) animal model of MS has shown that exercise protects against demyelination, increases brain-derived neurotrophic factor (BDNF), and reduces myelin damage and axonal damage. Consistent with pre-clinical research, MS work in humans has shown increased BDNF and reduction in pro-inflammatory circulating cytokines (i.e., IL-22) in those who exercised for 24 weeks versus those who maintained a sedentary lifestyle over the same period of time. In preliminary MS work from our group, 12 weeks of aerobic exercise resulted in increased hippocampal volume and hippocampal functional connectivity. Exercise is being considered as a candidate disease-modifying treatment. However, exercise is only beneficial if people do it. Despite the preponderance of evidence for exercise's salutary effects, many MS patients are deterred by overheating and exhaustion brought about by exercise. And while there is good evidence for the long-term safety profile of exercise in MS, many patients are put off by short-term discomforts, despite being physically capable of exercising.

Exercise causes overheating in people with MS. In healthy people, exercise triggers the conversion of metabolic to mechanical energy, resulting in the liberation of approximately 30-70% of the total energy as heat, which causes an increase in core body temperature. As core body temperature increases, exercise performance worsens. Exercise in persons with MS also raises body temperature, and heat-related MS symptoms increase following exercise. This is consistent with Uhthoff's phenomenon: the well-known deleterious impact of heat exposure and exercise for persons with MS. The investigators recently added an essential piece to this puzzle, reporting for the very first time that persons with relapsing-remitting MS (RRMS) have elevated body temperature even before being exposed to heat or exercising (i.e., at rest) relative to healthy controls. Importantly, this elevation in body temperature is clinically meaningful as warmer resting body temperature is linked to worse fatigue in patients with RRMS.Not only does this finding represent a paradigm shift in the conceptualization of heat sensitivity / heat exposure in persons with MS, but it highlights the additional burden of exercise-induced heat for people who are already warmer before exercise begins. Exercise increases body temperature in everyone; however, it was recently reported that only for persons with MS (compared to healthy controls) is exercise-induced increase in body temperature linked to exhaustion. Elevated body temperature at rest in persons with RRMS may be a key reason for this, and may also point to cooling as an effective treatment.

Cooling treatments are effective for people with MS. Elevated body temperature and its link to worse fatigue in RRMS patients aligns with positive results of several non-exercise trials of cooling treatments for reducing fatigue in MS patients none of which considered or targeted endogenously elevated body temperature. Aligned with this is evidence showing that cooling treatments administered to MS patients prior to or during exercise improve performance and reduce exhaustion. For example, in one study, ten MS patients used a hand-cooling chamber while walking on a treadmill: subjects kept one hand in the airtight device, a rigid chamber suspended by a bungee cord from above the treadmill throughout exercise. Cooling resulted in 33% increased exercise duration in the MS patients who kept their hand in the chamber. These findings support a beneficial impact of cooling during exercise, although these methods may be difficult to replicate / standardize, and implement clinically. In other work, whole-body precooling with a cooling vest and cap was used to successfully decrease perceived exertion during exercise. Yet another method of cooling via immersion in a cold water bath prior to exercise was found to reduce perceived exertion during exercise. By way of mechanism, Marino explained the heat-fatigue link in MS by proposing heat reaction blockade of action potentials in demyelinated neurons (i.e., frequency-dependent conduction block), noting that when demyelination is present, only a small increase in temperature (e.g., the amount induced by exercise) is necessary to completely block action potentials. This is consistent with seminal work in the giant squid axon demonstrating the disruption of action potentials in the presence of small, incremental increases in exogenous heat, ultimately resulting in reversible 'heat block' (cessation of neuronal conduction). An encouraging observation was that all effects of warming were completely reversible in this experimental model.

Cooling during exercise is an effective treatment for persons with RRMS. Taken together, the evidence supports cooling treatments as an effective means of improving exercise performance in patients with MS, although notably, no prior exercise study in MS has considered elevated core resting body temperature. Note that the finding of elevated body temperature was specific to RRMS; prior exercise cooling studies did not restrict their selection criteria to the relapsing-remitting phenotype. By doing so in the current proposal, the investigators expect to reveal a larger effect of cooling since relapsing-remitting MS patients with elevated body temperature at rest are most likely to experience exercise-induced fatigue (and are therefore most in need of effective cooling treatment). Prior methods of experimental cooling are cumbersome (e.g., cooling garments, immersion in a cool bath prior to exercise, insertion of one hand into a vacuum cooling chamber during exercise), thereby limiting replication and standardization for research use, and restricting practicality for clinical use. Here, the investigators propose to test the effectiveness of an oral antipyretic taken before exercise (i.e., administered 1-hour prior to exercise in order to reach peak serum concentration). Work in healthy adults has shown that antipyretic administration before exercise reduces body temperature during strenuous exercise in a hot environment, and improves performance (i.e., increases time-to-exhaustion). Aspirin (acetylsalicylic acid, ASA) has been selected, as it is shown to effectively reduce fatigue in prior non-exercise trials in MS (none of which considered aspirin's antipyretic mechanism of action as the key factor underlying treatment efficacy).

ELIGIBILITY:
Inclusion Criteria:

* RRMS
* self report of overheating during exercise
* low physical disability (EDSS total score 4.5 or less); fully ambulatory without aid
* exacerbation-free (and no use of corticosteroids) for 6 weeks prior
* BMI 35 or lower

Exclusion Criteria:

* uncontrolled hypertension or vascular disease of the legs
* current medications for heart or blood pressure problem
* prior history of head injury, stroke, or other neurological disease/disorder
* currently taking antipyretics or pain medication daily
* presence of major depressive disorder or other psychiatric diagnosis
* formally diagnosed sleep disorder
* pulmonary disease, heart disease or other heart problem
* diabetes mellitus or problem with blood sugar levels
* lower body weakness or reliance on supportive devices for walking (as indicated through EDSS)
* counter indications to aspirin use: history of confirmed peptic ulcer, gastrointestinal or sever gynecological bleeding; tarry stool or fecal occult blood; syndrome of asthma, rhinitis or nasal polyps

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01-13 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2017-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Leavitt, PhD, Principal Investigator — Assistant Professor of Neuropsychology
Locations (1):
- Columbia University Medical Center, MS Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Acetylsalicylic Acid at 1st Visit Then Placebo at 2nd Visit: Within-subjects design
  Participant is administered acetylsalicylic acid, an intervention to improve exercise performance (i.e., increase time to exhaustion) one hour prior to exercise.
  Acetylsalicylic acid: 650 mg dose of acetylsalicylic acid is administered in a capsule one hour prior to exercise
  Placebo Oral capsule: Placebo capsule is administered one hour prior to exercise
  First intervention: 1 day; washout period: 1 week; second intervention: 1 day
- Placebo at 1st Visit Then Acetylsalicylic Acid at 2nd Visit: Within-subjects design
  Participant is administered placebo one hour prior to exercise.
  Acetylsalicylic acid: 650 mg dose of acetylsalicylic acid is administered in a capsule one hour prior to exercise
  Placebo Oral capsule: Placebo capsule is administered one hour prior to exercise
  First intervention: 1 day; washout period: 1 week; second intervention: 1 day
Period: Overall Study
Arm/Group | Acetylsalicylic Acid at 1st Visit Then Placebo at 2nd Visit | Placebo at 1st Visit Then Acetylsalicylic Acid at 2nd Visit
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Because this was a within-subject design, participants received both drug and placebo, albeit at randomized visits. Therefore, all 12 analyzed participants were included in both trials.
Groups:
- Acetylsalicylic Acid at 1st Visit, Then Placebo at 2nd Visit: Participant is administered acetylsalicylic acid, an intervention to improve exercise performance (i.e., increase time to exhaustion) one hour prior to exercise.
  Acetylsalicylic acid: 650 mg dose of acetylsalicylic acid is administered in a capsule one hour prior to exercise
  Placebo Oral capsule: Placebo capsule is administered one hour prior to exercise
- Placebo at 1st Visit, Then Acetylsalicylic Acid at 2nd Visit: Participant is administered placebo one hour prior to exercise.
  Acetylsalicylic acid: 650 mg dose of acetylsalicylic acid is administered in a capsule one hour prior to exercise
  Placebo Oral capsule: Placebo capsule is administered one hour prior to exercise
- Total: Total of all reporting groups
Arm/Group | Acetylsalicylic Acid at 1st Visit, Then Placebo at 2nd Visit | Placebo at 1st Visit, Then Acetylsalicylic Acid at 2nd Visit | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  Overall Participants: <=18 years | 0 | 0 | 0
  Overall Participants: Between 18 and 65 years | 6 | 6 | 12
  Overall Participants: >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 2 | 2 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 6 | 12
Self-report heat-sensitivity during exercise [Count of Participants; unit: Participants] | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Time to Exhaustion
Description: The measure of interest is the length of time (in seconds) spent exercising at each session. This time has no pre-set upper limit, i.e. patients are free to exercise as long as they wish. This means that the time will not be censored. However, please note that healthy adults' time to exhaustion is approximately 12 minutes.
Time Frame: ASA's effect will be assessed from date of randomization until cessation of exercise test at each of two study visits to be completed within a 14-day period.
Population: All participants were recruited from the Columbia MS Center for Research and Treatment in New York, New York.
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Acetylsalicylic Acid: Participant is administered acetylsalicylic acid, an intervention to improve exercise performance (i.e., increase time to exhaustion) one hour prior to exercise.
  Acetylsalicylic acid: 650 mg dose of acetylsalicylic acid is administered in a capsule one hour prior to exercise
  Placebo Oral capsule: Placebo capsule is administered one hour prior to exercise
- Placebo Oral Capsule: Participant is administered placebo one hour prior to exercise.
  Acetylsalicylic acid: 650 mg dose of acetylsalicylic acid is administered in a capsule one hour prior to exercise
  Placebo Oral capsule: Placebo capsule is administered one hour prior to exercise
Arm/Group | Acetylsalicylic Acid | Placebo Oral Capsule
Number analyzed (Participants) | 12 | 12
seconds | 568 (150) | 552 (152)

2. Secondary Outcome: Exercise-induced Body Temperature Increase
Description: Measure of interest is increase in body temperature from pre- to post-exercise test in each treatment condition (ASA vs. placebo)
Time Frame: Effect of treatment on body temperature in a single session (i.e., pre- to post- exercise test) to be completed within a 14-day period
Population: subsample of people who self- identified as heat-sensitive during exercise (n=8)
Measure: Mean (Standard Deviation); unit: degrees Fahrenheit
Groups:
- Acetylsalicylic Acid: 650 mg dose of acetylsalicylic acid is administered in a capsule one hour prior to exercise
- Placebo Oral Capsule: Placebo capsule is administered one hour prior to exercise
Arm/Group | Acetylsalicylic Acid | Placebo Oral Capsule
Number analyzed (Participants) | 8 | 8
degrees Fahrenheit | 0.41 (0.55) | 0.88 (0.63)

ADVERSE EVENTS:
Time Frame: Adverse Event (AE) data were collected at any point during the study in which an AE arose: 2-3 weeks time for each participant
Arm/Group | Acetylsalicylic Acid | Placebo Oral Capsule
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
Small planned sample size in this pilot warrants follow-up replication in larger sample.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-01-30): https://cdn.clinicaltrials.gov/large-docs/46/NCT03051646/Prot_SAP_000.pdf
  • Informed Consent Form (2016-12-29): https://cdn.clinicaltrials.gov/large-docs/46/NCT03051646/ICF_001.pdf